CLINICAL TRIAL: NCT01744587
Title: Study of Epstein-Barr Virus Reactivation and the Effect of Dietary Supplement Epigallocatechin Gallate (EGCG) on Virus Reactivation in Remission Patients With Nasopharyngeal Carcinoma - A Randomized Trial
Brief Title: Epstein-Barr Virus Reactivation and the Effect of EGCG on Virus Reactivation in Remission Patients
Acronym: NPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Mackay Memorial Hospital (Other); Taichung Veterans General Hospital (Other); National Cheng-Kung University Hospital (Other); Chang Gung Memorial Hospital (Other); China Medical University Hospital (Other); National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: T2312
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: NPC
Keywords: EBV; EGCG
MeSH Terms: interventions — epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo qd (2# bid) for 3 years
  Interventions: Dietary Supplement: Placebo
- Epigallocatechin Gallate (EGCG) (Experimental): EGCG 600 mg qd (2# bid) for 3 years
  Interventions: Other: Epigallocatechin Gallate (EGCG)

INTERVENTIONS:
Other: Epigallocatechin Gallate (EGCG) — EGCG 600 mg per day will be provided to the test group.Four capsules will be taken daily (2# bid) by the test individuals.
  Other Names: EGCHAC-purified EGCG 90% capsules
  Arms: Epigallocatechin Gallate (EGCG)
Dietary Supplement: Placebo — Placebo qd (2# bid) for 3 years
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the EBV reactivation rate in post-radiation and remission NPC patients, evaluate the safety and tolerance of EGCG and analyze the observational correlation between EBV reactivation and clinical outcome.

DETAILED DESCRIPTION:
Patients with pathologically proven NPC, stage II-IVB and finishing curative RT ≧70 Gy within 6 months (± induction/concurrent/adjuvant chemotherapy) will be candidates for this study. Before entry, 8 CC venous blood will be obtained for EBV DNA and antibody screen tests after patient's consent. Those who have undetectable plasma EBV DNA (0 copy/ml) and fulfilled with all inclusion and exclusion criteria will be registered.

Routine re-staging work-ups after RT should show no active lesion in nasopharynx, neck and distant organs. Re-staging survey should include nasopharyngoscope, pEBV DNA assay, CBC, platelet count, renal and liver function tests, CXR, abdominal sonography or CT scan, whole body bone scan, MRI or CT scan of the head and neck region.

Within one week after finishing registration, EGCG or placebo should be started. A blood sample before taking EGCG/placebo will be collected for antibodies test and pEBV DNA assay.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven NPC.
* 2010 AJCC stage II-IVB.
* Age ≧ 20 years old.
* Performance status of ECOG ≦ 2.
* Finished RT ≧66 Gy within 6 months (± induction/concurrent/adjuvant chemotherapy).
* Clinical complete remission by re-staging work-ups within 3 months before entry.
* Plasma EBV DNA = 0 copy/ml within 4 weeks before entry.
* Adequate liver, renal, and bone marrow function:Serum total bilirubin level ≦ 2.5 mg/dl. Serum creatinine ≦ 1.6 mg/dl. WBC ≧ 3,000/ul. Platelet count ≧ 100,000/ul.
* No intake of EGCG or similar dietary supplements.
* Signed informed consent.
* No further anti-cancer treatment.

Exclusion Criteria:

* Occurrence of locoregional recurrence or distant metastasis.
* Inadequate RT or finishing RT > 6 months.
* Not complete remission by re-staging work-ups within 3 months before entry.
* Plasma EBV DNA > 0 copy/ml within 4 weeks before entry.
* Intake of EGCG or similar dietary supplements during recent 3 months.
* Severe cardiopulmonary diseases (unstable angina and/or congestive heart failure or peripheral vascular disease requiring hospitalization within the last 12 months; chronic obstructive pulmonary disease exacerbation other respiratory illness requiring hospitalization) or clinically significant psychiatric disorders.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
EBV reactivation rates between EGCG and placebo group | every 3 months for the first 3 years and every 6 months thereafter for antibodies tests and pEBV DNA assay (total 5 years)
  Reactivation of EBV is defined as
  1.Antibody against EBV VCA: The IgA antibody titers will be detected by a commercial EBV VCA ELISA kit (RE 562 71, Immuno-Biological Laboratories, Germany) Patient's serum with anti-EBV VCA greater than 10U/ml will be considered as reactivation of EBV.

SECONDARY OUTCOMES:
Correlation between EBV reactivation and OS/RFS | q 3 months for first 3 years and q 6 months for the
  Observational analysis of the correlation between EBV reactivation and clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Tsang Wu Liu, MD, Study Director — Taiwan Cooperative Oncology Group, National Health Research Institutes; Jin Ch Lin, MD PHD, Principal Investigator — Taichung Veterans General Hospital; Jen Ya Chen, PHD, Principal Investigator — National Institute of Cancer Research, National Health Research Institutes
Locations (1):
- Taiwan Cooperative Oncology Group, National Health Research Institutes, Zhunan, Miaoli, Taiwan